CLINICAL TRIAL: NCT05304143
Title: Efficacy of Immersive Entertainement Glasses in Magnetic Resonance Imaging to Reduce Claustrofobia: Clinical Control Trial
Brief Title: Efficacy of Immersive Entertainement Glasses in Magnetic Resonance Imaging (MRI)
Acronym: Claustro-VIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P/21-095
Record Dates: First submitted 2021-07-29; First posted 2022-03-31 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Claustrophobia; Magnetic Resonance Imaging (MRI)
Keywords: Immersive Entertainment Reality; Claustrophobia; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Claustrophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality intervention group (Experimental): The exploration in the intervention group will be carried out with virtual reality glasses compatible with the magnetic resonance imaging equipment.
  Interventions: Other: Virtual Immersive Reality Glasses
- Conventional nurse support (Active Comparator): The exploration in the control group will be carried out with the standard procedure for claustrophobic patients that includes close nursing support.
  Interventions: Other: Conventional nurse support

INTERVENTIONS:
Other: Virtual Immersive Reality Glasses — The day of the examination, the patient will go to the MRI room and he will be fitted with virtual reality glasses compatible with the MRI equipment. The patient will visualize relaxing contents in open spaces with music and verbal instructions during all the procedure. The contents will be previously validated by the clinical psychologist of the center with experience in this regard.
  During the test, the patient's heart rate will be monitored.
  Arms: Virtual Reality intervention group
Other: Conventional nurse support — Patients will be treated using the usual support technique to reduce anxiety in the Diagnostic Imaging service
  Arms: Conventional nurse support

SUMMARY:
Background: Claustrophobia is the most common type of specific phobia, and in the context of performing an MRI, it leads to premature completion of the test or a sedation. According to some authors, 1,6% of the patients terminated the test prematurely due to claustrophobia, and, in addition, 3.8% underwent conscious sedation. These procedures increase the risk of complications, and the cost of care. The use of anxiolytics is an option to reduce anxiety, but these drugs carry the possibility of suffering adverse effects, and the fact that patients cannot drive home when the MRI is finished. For these reasons, it is especially relevant to determine which non-pharmacological interventions are most effective, and among them, the use of Immersive Entertainment Glasses is a low-interventionist option that can help to overcome fear of the test.

Objective: To determine the effectiveness of Immersive Entertainment Glasses in the success of the performance of an MRI and in the reduction of anxiety levels, in patients who express having claustrophobia.

Methodology:

Design: Clinical trial with intervention and control group. Participants: patients who define themselves as claustrophobic and should have an MRI. The sample will be made up of 206 individuals, divided between an intervention group and a control group. expecting a 20% difference between the success of the test of the control and intervention group subjects.

People who meet the inclusion criteria will be distributed into the control or intervention group. The intervention group will use the Immersive Entertainment Glasses to perform the MRI and the control group will have the support of the nurse through educational techniques.

Expected results: the success rate in performing MRIs is expected to increase by 20%, thanks to the use of Immersive Entertainment Glasses.

Expected duration: 12 months, or until obtaining the expected sample.

DETAILED DESCRIPTION:
INTRODUCTION According to the Diagnostic and Statistical Manual of Mental Disorders (DSM V), there are many categories of anxiety disorders. The specific phobias are a type of disorder where there is an extreme fear of people, objects, or specific situations. Among the most common symptoms are physical and emotional ones. Physical symptoms may include, but are not limited to, shortness of breath, trembling, sweating, tachycardia, dry mouth, and chest pain. The most frequent emotional symptoms are feeling overwhelmed by anxiety or fear, presenting fear of losing control, needing to leave the place that causes anxiety and understanding that it is an irrational fear but not being able to avoid it. According to some authors, the specific disorders in the Korean population are between 5.2% and 4.2%.

Among the different phobias, claustrophobia is the most common. This is a situational phobia and consists of an irrational fear that occurs when the person is in closed spaces such as an elevator, a tunnel, or some radiological test equipment such as an MRI. The person has an intense and irrational fear of being confined in a small space and not being able to escape.

This situation has an implication from the point of view of public health because these people are sometimes unable to undergo an MRI since, in addition, they must be about 30 minutes still in a small space. Therefore, this type of disorder leads on numerous occasions to the cancellation of the test, or to a premature termination, causing damage to the patient's health since, either the MRI is not performed, or they must undergo sedation or anesthesia.

Magnetic resonance imaging is very useful in the detection and characterization of lesions. Some authors state that 37% of people who undergo an MRI have moderate to intense levels of anxiety. The prevalence of claustrophobia in the population is between 7.7% and 12.5%, although the frequency is higher among the female sex Approximately 1% of the population that requires an MRI rejects its performance or terminates it prematurely due to claustrophobia. Some researchers claim that 1.6% of patients finished the test prematurely due to claustrophobia, and, in addition, 3.8% underwent conscious sedation. These procedures increase the risk of complications, and in addition they increase the cost.

The most common therapy to treat claustrophobia is cognitive behavioral therapy, with gradual exposure to closed or narrow spaces being the most widespread treatment.

The use of some drugs, such as anxiolytics, is an option to reduce anxiety before imaging procedures. However, these drugs introduce some drawbacks such as all their adverse effects. For this reason, it is especially important to determine which are the non-pharmacological interventions that are most effective.

In this context, new technologies such as Immersive Entertainment Glasses (IEG) allow patients to feel immersed in another reality, open and relaxing, which helps them overcome this situation. Some studies state that these strategies are useful for reducing the symptoms produced by claustrophobia. In addition, the use of virtual reality glasses as a distraction element is more effective than music therapy against claustrophobia.

JUSTIFICATION Currently, at the Hospital Universitari Mútua de Terrassa, patients who report claustrophobia or fear of undergoing the test due to feeling confined or being unable to be inside the magnet, are referred to an open MRI scan at another health center. This means that patients must go to a private health center and undergo a test of inferior technical quality, since the open magnets have a low magnetic field, which limits the quality of the studies. The implementation of techniques that help reduce claustrophobia can avoid some sedation or anesthesia and, in addition, some people will be able to perform the test without pharmacological assistance and with higher quality images, which will improve their diagnosis.

HYPOTHESIS AND OBJECTIVES MAIN OBJECTIVE To identify the effectiveness of the use of IEG during the performance of an MRI in patients who express claustrophobia.

SPECIFIC OBJECTIVES

1. Assess the quality of the images obtained from the studies carried out in the intervention group (IG) and in the control group (CG)
2. Determine the number of tests that ended prematurely in the intervention group (IG) and in the control group (CG)
3. To identify the levels of state-anxiety and trait-anxiety through the State Trait Anxiety Inventory questionnaire (A/E and A/R) before and after the resonance in the control group (CG) and the intervention group (IG)
4. Compare the heart rate (HR) of the patients during the test with respect to the before value
5. Assess the satisfaction of patients in the intervention group in relation to the use of IEG.

HYPOTHESIS Implementing the use of IEG (Cinema Vision®, General Electric), with distracting content, in magnetic resonance imaging studies in patients who report fear of closed spaces, will reduce state-anxiety values, and increase the number of patients who will undergo the test successfully in at least 20%, compared to the previous situation.

MATERIAL AND METHODS

Design:

Clinical trial with random assignment of patients to a control group and an intervention group.

The study will be carried out at the facilities of the Diagnostic Imaging Department of the Hospital Universitari Mútua de Terrassa with a General Electric (GE) 1.5 Tesla MRI. For the IG, all examinations will be performed on an MRI to which the IEG have been added, and for the CG they will be performed on the same MRI or on another with the same characteristics without the installation of IEG.

Study population:

Patients who are defined as claustrophobic and who should undergo an MRI at the Hospital Universitari Mútua de Terrassa (HUMT).

Sample size and justification:

During 2019, a total of 252 patients were referred to another center to perform an MRI for referring claustrophobia. The sample will consist of 206 individuals, divided between an IG and a CG. With an alpha risk of 0.05 and a beta risk of less than 0.2, in unilateral contrast, with 103 subjects in each group, expecting a difference of 20% between the success of performing the test of the subjects of the control group and intervention. The estimated loss rate has been established at 0 because possible withdrawls will be exchanged with other participants.

The selection of patients will be carried out consecutively in all the patients who are requested to have an MRI and who define themselves as claustrophobic and relate to the Diagnostic Imaging Department of HUMT and will be distributed randomly in the two groups.

Data collection and intervention procedure Requests that arrive at the External Referral Service due to claustrophobia will be sent to the Diagnostic Imaging Department to be included in the study. Potential participants will first be contacted by phone to find out if they meet the study inclusion criteria and will be offered to participate in the study. These patients would have been referred for open MRI or sedation. The patient will receive an information sheet explaining the purpose of the study and an informed consent sheet. All patients who meet the inclusion criteria and sign the informed consent will be included in the study. The patient can revoke consent at any time. These patients will be scheduled on separate days from the rest to perform the test with the intervention of IEG or with professional support.

To measure anxiety levels, the State-Trait Anxiety Questionnaire (STAI, State-Trait Anxiety Inventory Self Evaluation Questionnaire), will be used before the test, which will allow to differentiate between anxiety as a personality trait or as a state caused by the test (STAI-E and STAI-R). After the MRI, the STAI-E will be administered again, to compare the state of anxiety pre-post examination. The anxiety-state scale (A/E) is used to determine the levels of anxiety induced by experimental procedures with tension or stress load. A/E scores increase in response to different types of stress and decrease with relaxation techniques. This questionnaire is one of the classic measures to assess anxiety and is considered one of the references.

Patients will be appointed to the CG or IG alternately and consecutively in the inclusion process. On the day of the examination, the patient will go to the MRI room and, if they belong to the IG, they will be fitted with IEG compatible with the MRI. The patient will view the content chosen by him or her during the test. Relaxing content will be offered with music and verbal instructions. The contents will be previously validated by the center's clinical psychologist with experience in this matter.

During the test, the patient's heart rate will be monitored. Once the examination has been carried out, patient satisfaction will be assessed using an ad hoc questionnaire.

Likewise, the quality of the images will be analyzed, and the data collected will be recorded in a specific database for this study.

A pilot test will be carried out with 15 patients to detect possible limitations or improvements.

Study variables:

Independent variable: type of intervention performed, that is, IEG glasses or the usual procedure.

Dependent variables:

* Percentage of patients who complete the MRI, that is, percentage of success.
* In addition, the quality of the images of the studies carried out will be assessed using a Likert scale (with values between 1 and 4), where value 1 is very low quality and non-assessable studies and value 4 is the expected maximum. This parameter will be assessed by the nurse performing the test.
* Variables regarding the IEG: in terms of satisfaction, patients will be asked if they would recommend the experience to other people, if they think that the IEG have helped them to carry out the test and if they have found it pleasant. This will be assessed through a Likert scale with 10 values, where 0 corresponds to a low assessment and 10 to the highest score.
* Other variables: anxiety values before and after the test (STAI pre-post RM), heart rate at the beginning and end.

Control variables:

* Sociodemographic variables: initials of the patient's name and surnames, medical record number, age, sex.
* Variables regarding the test: diagnosis that caused the inquiry, part of the body explored, if it has a previous MRI, and if so, if it was an open or closed MRI, if parts of the test had to be repeated, or if the complete MRI could be performed (successfully).

Sources of information and obtaining information The sources of information include the data provided by the patient and his or her clinical history, as well as the data that will be collected during the development of the study.

* Ad hoc questionnaire to collect the variables described
* STAI Questionnaire -State Trait Anxiety Inventory

Statistical analysis:

For the statistical analysis, the statistical program SPSS for Windows will be used. First, a descriptive study of the sample will be carried out using measures of central tendency and dispersion. The results of the sociodemographic and baseline anxiety variables of the participants in both groups will be compared to assess their comparability. The association of the variables will be studied using the Chi2 and Student's t tests, and the anxiety and heart rate variables will be analyzed using the McNemar test for proportions with paired data.

Study limitations:

The patient's anxiety to know the result of the test can influence the anxiety-state values and interfere with the concern that the patient presents for the diagnostic imaging test.

Another possible limitation may be that the difference between patients who receive support through educational measures and EG is less than the 20% estimated according to the literature, and therefore, the sample should be larger.

If the CG presents higher levels of anxiety than the IG, this will also imply a limitation of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with self-reported fear of enclosed spaces
* Patients with fear of having an MRI

Exclusion Criteria:

* Patients who must undergo a sustained breathing exploration during the test
* Patients who have a contraindicated MRI
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Succes in the performance of an MRI | One hour
  Number of patients that will finish the MRI
Anxiety reduction | One hour
  Decrease of the levels of anxiety measured with the State Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Image quality | Half an hour
  The images will be evaluated by the nurse in a Likert Scale
Failed MRI | One hour
  Number of unfinished exams
Patient satisfaction | One hour
  Satisfaction measured with a ad hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Díaz Membrives, PhD, Principal Investigator — Supervisor of Imaging Diagnostics
Locations (1):
- Mútua de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Carpenter JK, Moskow DM, Hofmann SG. Enhanced Mental Reinstatement of Exposure to Improve Extinction Generalization: A Study on Claustrophobia and MRI Fear. Behav Ther. 2023 Jan;54(1):156-169. doi: 10.1016/j.beth.2022.08.002. Epub 2022 Aug 13. PMID 36608973
- [Background] Brown RKJ, Petty S, O'Malley S, Stojanovska J, Davenport MS, Kazerooni EA, Fessahazion D. Virtual Reality Tool Simulates MRI Experience. Tomography. 2018 Sep;4(3):95-98. doi: 10.18383/j.tom.2018.00023. PMID 30320208
- [Background] Pull CB. Recent trends in the study of specific phobias. Curr Opin Psychiatry. 2008 Jan;21(1):43-50. doi: 10.1097/YCO.0b013e3282f30086. PMID 18281840
- [Background] Rahani VK, Vard A, Najafi M. Claustrophobia Game: Design and Development of a New Virtual Reality Game for Treatment of Claustrophobia. J Med Signals Sens. 2018 Oct-Dec;8(4):231-237. doi: 10.4103/jmss.JMSS_27_18. PMID 30603615
- [Background] Tugwell JR, Goulden N, Mullins P. Alleviating anxiety in patients prior to MRI: A pilot single-centre single-blinded randomised controlled trial to compare video demonstration or telephone conversation with a radiographer versus routine intervention. Radiography (Lond). 2018 May;24(2):122-129. doi: 10.1016/j.radi.2017.10.001. Epub 2017 Oct 31. PMID 29605108
- [Background] Garcia-Palacios A, Hoffman HG, Richards TR, Seibel EJ, Sharar SR. Use of virtual reality distraction to reduce claustrophobia symptoms during a mock magnetic resonance imaging brain scan: a case report. Cyberpsychol Behav. 2007 Jun;10(3):485-8. doi: 10.1089/cpb.2006.9926. PMID 17594277
- [Background] King S, Woodley J, Walsh N. A systematic review of non-pharmacologic interventions to reduce anxiety in adults in advance of diagnostic imaging procedures. Radiography (Lond). 2021 May;27(2):688-697. doi: 10.1016/j.radi.2020.09.018. Epub 2020 Oct 4. PMID 33028496
- [Background] Spielberger CD Lushene PR, Jacobs GA. GRL. Manual for the State-Trait Anxiety Inventory. Consult Psychol Press. 1983.
- [Background] Vadakkan C, Siddiqui W. Claustrophobia. 2023 Feb 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK542327/ PMID 31194467
- [Derived] Diaz-Membrives M, Garrido-Ribas I, Caro-Benito C, Font-Cabrera C, Monistrol O. Claustrophobia in magnetic resonance imaging: A randomised controlled trial of immersive entertainment glasses. Radiography (Lond). 2026 Jan 3;32(2):103318. doi: 10.1016/j.radi.2025.103318. Online ahead of print. PMID 41485316